CLINICAL TRIAL: NCT02709200
Title: Effect of Dexmedetomidine on Pacemaker Function Following Cardiac Surgery
Status: Withdrawn | Type: Observational
Why Stopped: Unable to enroll subjects.
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chief, Department of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Other Study IDs: IRB13-00127
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dexmedetomidine: Patients that received dexmedetomidine during open heart surgery.
  Interventions: Drug: Dexmedetomidine
- No dexmedetomidine: Patients that didn't receive dexmedetomidine during open heart surgery.

INTERVENTIONS:
Drug: Dexmedetomidine
  Other Names: Precedex
  Groups: Dexmedetomidine

SUMMARY:
This is a prospective study looking at the effects of dexmedetomidine on pacemaker function in patients who have surgery for congenital heart disease utilizing cardiopulmonary bypass (CBP). For the purpose of the study, no change in intraoperative care will be dictated. The use of dexmedetomidine will be left up to the discretion of the treating physicians. The study will involve only the collection of data regarding the amplitude required to capture and specific demographics and intraoperative features including cross clamp time, time on CPB, and vasoactive agents that were and are being administered. In addition to these data, it will be noted whether dexmedetomdine was used or not and whether it is being administered on arrival to the CTICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients with temporary surface pacemaker leads following surgery for congenital heart disease.

Exclusion Criteria:

* Patients with single ventricle anatomy
* Patients receiving epinephrine
* Infants less than 6 months of age

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Congenital heart disease patients having open heart surgery.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Amplitude | Baseline
  The impulse required to elicit atrial or ventricle capture (contraction) of the surface electrode of a temporary postoperative pacemaker.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No